CLINICAL TRIAL: NCT02245373
Title: Cost-effectiveness of a Non-Pharmacological Treatment (Active Monitoring) vs. a Pharmacological Treatment for Major Depression in Primary Care. INFAP Study.
Brief Title: Cost-effectiveness of a Non-Pharmacological Treatment (Active Monitoring) vs. a Pharmacological Treatment for Major Depression in Primary Care.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Other Study IDs: Infap
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Mild to Moderate Depression.
Keywords: Depression; Primary Care; Cost-effectiveness; Pharmacological treatment; Watchful-waiting or Active Monitoring.
MeSH Terms: conditions — Depression | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

GROUPS / COHORTS (2):
- Antidepressants: Naturalistic assignment: Patients whose physician decides to indicate antidepressants.
  Interventions: Drug: Antidepressants
- Active Monitoring: Naturalistic assignment: Patients whose physician considers starting an Active Monitoring intervention.
  Interventions: Other: Active Monitoring

INTERVENTIONS:
Drug: Antidepressants
  Groups: Antidepressants
Other: Active Monitoring
  Groups: Active Monitoring

SUMMARY:
Major Depression (MD) is highly prevalent and has associated a high burden and economic costs. Mild levels of MD could be treated without antidepressants at Primary Care (PC).

Main objectives: 1) To calculate the cost-effectiveness of active monitoring (recommended by NICE) vs pharmacological antidepressant treatment to treat mild MD at PC level.

Methods: 300 patients (≥18 years) with MD (diagnosed by the GP) will be recruited at the PC center. Depending on the level of symptoms, the GP will choose between: A) Active Monitoring (n=150) and B) pharmacological treatment (n=150).

Patients will be followed-up for one year and data will be collected at baseline, 6 and 12 months. Severity will be assessed by Patient Health Questionnaire (PHQ-9), quality of life with the EuroQoL-5D (5 health dimensions), and the use of services with an adapted version of the Client Service Receipt Inventory (including lost productivity).

Cost-effectiveness and cost-utility analysis will be calculated and 5000 bootstrapping replications will be conducted to asses uncertainty. Cost-acceptability curves will be done using two perspectives: the National Health Service perspective and the Societal perspective.

The Propensity Score technique will minimize the absence of randomization, matching cases from both treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose GP considers to have major depression. The indication of pharmacological or non-pharmacological treatment will be based strictly on the clinical judgment of the physician.
2. Adults (≥18 years)
3. Informed consent signed by the physician and the patient to participate in the study.

Exclusion Criteria:

1. Use of antidepressant drugs during the previous 60 days to inclusion date.
2. Alcohol or other toxic abuse.
3. Psychosis or bipolar disorder identified in the psychiatric interview
4. Use in the last 6 months of antipsychotic drugs, lithium or antiepileptic
5. Health status (pregnancy) and / or disease and / or treatments that contraindicate the use of antidepressant drugs.
6. Terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients who suffer from major depression.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Compare the cost-effectiveness of active monitoring (standard treatment without antidepressants) vs antidepressants in mild major depression taking into account the severity and disability in Primary Care. The changes at Time Frame will be assessed. | At base Line, 6 months and 12 months.
  Measures: Severity of Depression (PHQ-9), Quality of life (EuroQol) and the use of services (Client Service Receipt Inventory, CSRI).

SECONDARY OUTCOMES:
1.Quality of life of patients with major depression who initiate treatment in Primary Care. | At base line, 6 months and 12 months.
2. Cost-utility of an antidepressant vs no treatment in mild Depression in Primary. | At base line, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Serrano, PhD, Principal Investigator — Fundació Sant Joan de Déu

REFERENCES:
- [Derived] Rubio-Valera M, Beneitez I, Penarrubia-Maria MT, Luciano JV, Mendive JM, McCrone P, Knapp M, Sabes-Figuera R, Kocyan K, Garcia-Campayo J, Serrano-Blanco A. Cost-effectiveness of active monitoring versus antidepressants for major depression in primary health care: a 12-month non-randomized controlled trial (INFAP study). BMC Psychiatry. 2015 Mar 31;15:63. doi: 10.1186/s12888-015-0448-3. PMID 25885818